CLINICAL TRIAL: NCT07125963
Title: Comparison of a Patient-Specific Proximal Segment Positioning Appliance and the Conventional Method in Sagittal Split Ramus Osteotomy
Brief Title: Patient-Specific vs. Conventional Positioning in Sagittal Split Ramus Osteotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sümer Münevveroğlu (Other)
Responsible Party: Sponsor-Investigator, Sümer Münevveroğlu, Assistant Professor, Medipol University
Organization: Medipol University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MEDIPOL-SSRO-001
Record Dates: First submitted 2025-07-29; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-01

CONDITIONS: Dentofacial Deformities
Keywords: Sagittal Split Ramus Osteotomy; Orthognathic Surgery; 3D Surgical Planning; Patient-Specific Guide; Proximal Segment Position
MeSH Terms: conditions — Dentofacial Deformities

STUDY DESIGN:
Intervention Model Description: This study uses a split-mouth crossover design. Each patient receives both interventions: a custom-made positioning appliance is applied to one side of the mandible, while the contralateral side is positioned using the conventional manual method. This intra-patient comparison allows direct assessment of positional accuracy and clinical effectiveness between the two techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom-made positioning appliance-assisted mandibular segment repositioning (Experimental): Patients receive a custom-made positioning appliance designed via STL-based planning and manufactured using 3D printing. The appliance is used to guide the proximal mandibular segment during sagittal split ramus osteotomy on one side of the mandible, aiming to improve positional accuracy.
  Interventions: Procedure: Custom-made positioning appliance-assisted mandibular segment repositioning
- Conventional Manual Positioning (Active Comparator): On the contralateral side of the mandible, the proximal segment is positioned manually by the surgeon using standard visual and tactile feedback during sagittal split ramus osteotomy, without a guiding appliance.
  Interventions: Procedure: Conventional Manual Positioning

INTERVENTIONS:
Procedure: Custom-made positioning appliance-assisted mandibular segment repositioning — A patient-specific surgical guide designed using STL-based digital planning in Blender and produced via 3D printing with biocompatible surgical resin (Formlabs SLA printer). Used to guide and stabilize the proximal mandibular segment during sagittal split ramus osteotomy.
  Arms: Custom-made positioning appliance-assisted mandibular segment repositioning
Procedure: Conventional Manual Positioning — The proximal mandibular segment is positioned manually by the surgeon based on visual and tactile feedback without the use of a positioning guide. This technique represents the standard method in sagittal split ramus osteotomy.
  Arms: Conventional Manual Positioning

SUMMARY:
This study aims to evaluate the clinical efficacy and positioning accuracy of a custom-made proximal segment positioning appliance designed for use in sagittal split ramus osteotomy (SSRO). The appliance is produced using STL-based digital planning and 3D printing technologies. In each patient, the appliance is applied to one side of the mandible while the contralateral side is positioned using the conventional manual method. This within-subject design enables direct comparison by eliminating inter-individual anatomical variability. The primary outcome is the accuracy of segment positioning, evaluated by 3D superimposition and deviation analysis of pre- and postoperative STL models. Secondary outcomes include surgical time, ease of use as rated by the surgeon, and postoperative temporomandibular joint symptoms. The study will enroll 30 adult patients undergoing SSRO or double-jaw surgery due to dentofacial deformities. The results are expected to provide high-level clinical evidence for the reliability of patient-specific appliances in orthognathic surgery.

DETAILED DESCRIPTION:
Sagittal split ramus osteotomy (SSRO) is a widely used orthognathic surgery technique to correct mandibular deformities. During SSRO, accurate positioning of the proximal segment is critical for ensuring temporomandibular joint (TMJ) health, symmetry, and long-term surgical stability. However, conventional positioning relies heavily on the surgeon's visual judgment and experience, which may lead to postoperative complications such as condylar displacement, facial asymmetry, and TMJ dysfunction.

This prospective, randomized clinical study introduces a patient-specific proximal segment positioning appliance developed through STL-based 3D design using Blender and printed with biocompatible surgical guide resin via a Formlabs SLA 3D printer. Each patient will undergo SSRO (with or without Le Fort I osteotomy), and the custom appliance will be used to guide the proximal segment on one mandibular side. The opposite side will be positioned conventionally, allowing intra-patient comparison.

Postoperative CBCT images will be obtained at 1 month and converted to STL format. These models will be aligned with preoperative plans using MeshLab software to evaluate linear and rotational deviations. Surgical time, ease of application, and TMJ symptoms will be documented. Statistical analysis will include paired t-tests or Wilcoxon signed-rank tests depending on data distribution.

This study will generate clinically meaningful data regarding the effectiveness and safety of patient-specific guides in mandibular segment positioning. The proposed method also holds commercialization potential and may reduce intraoperative variability and dependence on surgeon experience.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo bilateral sagittal split ramus osteotomy as part of orthognathic surgery
* Age ≥ 18 years
* Availability of preoperative and postoperative CT scans
* Consent to participate in the study

Exclusion Criteria:

* History of previous mandibular surgery
* Craniofacial syndromes or congenital deformities
* Incomplete radiological records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Deviation of the proximal mandibular segment from the preoperative plan | 1 Month Postoperatively
  The deviation between the actual postoperative position of the proximal mandibular segment and the virtually planned position will be measured in millimeters using superimposed STL files in MeshLab software. The mean deviation value will be compared between the custom-made positioning appliance-assisted method and conventional manual positioning to assess positional accuracy.

SECONDARY OUTCOMES:
Duration of Fixation After Split | Intraoperative
  The time required for fixation of the mandibular segments following sagittal split osteotomy will be recorded separately for each side. This period begins immediately after the osteotomy is completed and ends when rigid fixation is achieved. The recorded times will be compared between the custom-made positioning appliance-assisted method and the conventional manual method to evaluate potential differences in procedural efficiency.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Medipol Mega University Hospital, Istanbul, Bağcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and institutional policy restrictions regarding the sharing of de-identified clinical data.